CLINICAL TRIAL: NCT05813522
Title: Efficacy and Safety Analysis of Furmonertinib in Patients With Leptomeningeal Metastases Associated With EGFR Mutated NSCLC，Guiding by Cerebrospinal Fluid ctDNA Detection
Brief Title: Furmonertinib in Patients With Leptomeningeal Metastases Associated With EGFR Mutated NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHNFLM-IIT-01
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Leptomeningeal Metastases; EGFR mutations; Furmonertinib; ctDNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis | interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (Experimental): Furmonertinib 160mg po qd
  Interventions: Drug: Furmonertinib Mesilate Tablets

INTERVENTIONS:
Drug: Furmonertinib Mesilate Tablets — 160mg of Furmonertinib mesilate tablets (given as four 40mg tablets) administered orally once daily
  Other Names: AST2818

SUMMARY:
The goal of this clinical trial is to evaluate the clinical efficacy and safety of Furmonertinib in EGFR mutated NSCLC patients with leptomeningeal metastasis and to explore the feasibility of CSF ctDNA detection for efficacy evaluation. Participants will be treated with 160mg Furmonertinib daily and tumor evaluation will be performed every 6-8 weeks. The participants' blood and cerebrospinal fluid samples will be collected three times during the study for ctDNA detection.

DETAILED DESCRIPTION:
Advanced non-small cell lung cancer patients with leptomeningeal metastases tend to have a worse prognosis. Currently, no standard therapeutic regimen for LM has been established because of its rarity and heterogeneity. Targeted therapy is the primary treatment of patients with EGFRm of NSCLC. The drug concentration in cerebrospinal fluid is the key factors affecting the curative effect of intracranial metastatic lesions. The widespread application of EGFR-TKIs in clinical practice has significantly prolonged the survival period of patients with EGFR mutations, but the standard dose of first- and second-generation EGFR-TKIs show poor control of intracranial metastasis.Furmonertinib is a third-generation EGFR-TKI targeting both sensitising EGFR and EGFR T790M mutations. Phase 2 clinical study of furmonertinib revealed that furmonertinib was clinically effective with acceptable toxicity in patients with EGFR T790M mutated advanced NSCLC, including in patients with CNS metastases. At present, some study has found that the dynamic changes of EGFR in plasma ctDNA can be used to evaluate the prognosis of NSCLC patients. Some study has also observed that the copy number variations in CSF ctDNA of NSCLC patients with LM are related to the curative effect. Therefore, CSF ctDNA may become a new biomarker to assess the therapeutic effect of LM. This is a single-center, open, single-arm, exploratory phase 2 trial evaluating the clinical efficacy and safety of Furmonertinib in EGFR mutated NSCLC patients with leptomeningeal metastasis and to explore the feasibility of CSF ctDNA detection for efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures.
2. Age ≥18 years.
3. Newly diagnosed NSCLC patients with leptomeningeal metastases associated with EGFR activating mutant or patients who develop leptomeningeal metastases only after treatment with first- or second-generation of EGFR-TKIs.
4. LM diagnosis was based on the detection of malignant cells in the CSF. Patients with new neurological symptoms and signs or typical MRI findings, together with the EGFR mutations detected by CSF ctDNA, can also be enrolled even if CSF cytology is not positive.
5. Subjects may be eligible for or have had CNS shunt or Ommaya fluid reservoir implantation. Patients who do not meet the requirements should be able to cooperate with lumbar puncture.
6. ECOG performance status of 0 to 2.
7. Life expectancy ≥ 3 months.
8. Patients must have stable extracranial symptoms and have no CNS complications requiring urgent neurosurgical intervention for at least 4 weeks before study enrollment.
9. At least one measurable extracranial lesion as defined by RECIST 1.1.
10. Women of childbearing age (WOCBP) and male subjects should take effective contraception during the treatment and within 3 months after the end of treatment. WOCBP should be non-pregnant within 1 week prior to study enrollment.

Exclusion Criteria:

1. Previous or current treatment of any third-generation EGFR-TKI.
2. Previously treated with radiotherapy for central nervous system metastases.
3. A history of stroke within 6 months or pre-existing central nervous system damage which can interfere with neurological evaluation.
4. A history of chronic gastrointestinal disease or any other medical condition that would preclude adequate absorption of Furmonertinib.
5. Currently receiving (or unable to stop use at least 1 week prior to receiving the first dose of Furmonertinib) medications or herbal supplements known to be potent inhibitors or inducers of CYP3A4/5.
6. A history of previous or current tumors other than NSCLC, with the exception of radical non-melanoma skin cancer, carcinoma in situ of the cervix, benign prostate tumor/hypertrophy, or other cancers that have been radical and have no evidence of relapse for at least 5 years.
7. Past medical history of any kinds of interstitial lung disease or radiation pneumonitis.
8. Systemic antitumor therapy with other agents was planned before enrollment or during the duration of the study.
9. Major surgery procedure or significant traumatic injury within 2 weeks of the first dose of study treatment.
10. A history of hypersensitivity reactions to the study medicine.
11. Peripheral neuropathy,greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment.
12. Any evidence of severe or uncontrolled serosal effusion and systemic diseases, including uncontrolled hypertension, diabetes, cardiovascular disease, active bleeding diatheses and severe acute or chronic infections that require systemic treatment(including positive HbsAg or positive HCV antibodies or confirmed positive HIV test result).
13. Inadequate bone marrow reserve or organ function.
14. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial Progression-Free Survival (PFSi) | Assessed up to 12 months.
  PFSi is defined as the time from first dose of Furmonertinib in this study until the date of intracranial disease progression.
Overall Progression-Free Survival (PFSo) | Assessed up to 12 months.
  PFSo is defined as the time from first dose of Furmonertinib in this study until the date of disease progression.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Assessed up to 12 months.
  ORR is defined as the percentage of patients with a best response of CR (complete response) or PR (partial response).
Disease Control Rate (DCR) | Assessed up to 12 months.
  DCR is defined as the proportion of patients with a best overall, extracranial and CNS, respectively, response of confirmed CR, confirmed PR, or SD.
Overall Survival (OS) | Assessed up to 24 months.
  OS is defined as the time from the date of first dose of Furmonertinib in this study until death due to any cause.

OTHER OUTCOMES:
Adverse events/Serious adverse events | From signing ICF to 30 days after the end of treatment.
  Incidence of Adverse Events (AEs): Incidence, severity and seriousness of adverse events, incidence of serious adverse events (SAEs), which usually be graded by CTCAE v5.0 based on current clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehong Wang, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share participant data of the trial.